CLINICAL TRIAL: NCT02804321
Title: Plasma Aldosterone Levels and Atrial Fibrillation Reduction (ALDO-AF Study)
Acronym: ALDO-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A13-D37-VOL.18
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation; Aldosterone
Keywords: catheter ablation; galectin 3; ngal; aldosterone; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — aldosterone galectine 3 ngal
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmias with a constantly growing prevalence. Two main techniques are used today to restore sinus rhythm: electrical cardioversion and radiofrequency ablation.

Radiofrequency ablation has become a recognized and effective treatment of AF. Despite a relatively high success rate (about 80%), a substantial number of patients require a second procedure to obtain sinus rhythm. Many publications have led to the study of predictors of failure of this ablation factors (BMI, uncontrolled hypertension, size of the OG...) but to date no parameter is reliable and usable in daily practice.

It is the same for electrical cardioversion. Despite a relatively high immediate success rate of approximately 80%, a significant number of patient relapse arrhythmia in short and long term. Many publications have led to the study of predictive factors of failure (seniority and type of AF, uncontrolled hypertension, size of the OG, mitral valve disease...) but so far the results are disappointing.

In AF patients with heart disease underlying, it has been well demonstrated that the renin-angiotensin system (RAAS) was strongly activated. In addition, it is now well established that elevated plasma aldosterone as in primary hyperaldosteronism is associated with a significantly increased risk of occurrence of cardiovascular events. The high plasma concentrations were also highlighted in the acute phase of myocardial infarction, or heart failure and are associated with an increase in major cardiovascular event rate, especially arrhythmias. In some experimental models of heart failure, it has been demonstrated a suppression of the occurrence of spontaneous FA by an anti-aldosterone treatment. The arrhythmogenic effect of aldosterone has also been shown in animal models. All these results indicate a potential role of aldosterone in the genesis of an arrhythmogenic substrate and the FA.

The hypothesis of this study is that aldosterone plasma levels in pre-reduced patients is predictive of recurrence risk of atrial fibrillation or other supraventricular tachycardias (flutter or atrial tachycardia) after FA reduction, either in using a radiofrequency ablation or via electrical cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for atrial fibrillation cardioversion by radiofrequency ablation or electrical cardioversion
* scheduled hospitalisation or hospitalisation unrelated to cardiovascular events
* Age at least 18 years
* Clinically Stable (see criteria for non-inclusion)

Exclusion Criteria:

* Patient unstable defined as any cardiovascular event that occurred in the previous 30 days

These events are:

* hospitalisation for cardiovascular causes
* appearance or worsening of symptoms consistent with cardiac failure
* appearance or worsening symptoms of coronary

  * Patient refusing participation in the study
  * Patient unable to provide follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to all patients referred for atrial fibrillation cardioversion by radiofrequency ablation or electrical cardioversion, clinically stable, at Caen University Hospital, Pitié-Salpêtrière and Ambroise Paré clinic.
  These patients have a strict, rigorous and systematic follow after these cardioversion at 1, 3 and 6 months with routine ECG.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
recurrence of supraventricular tachycardia (atrial fibrillation, atrial flutter and atrial tachycardia) after atrial fibrillation reduction by radiofrequency ablation or electrical cardioversion. | 6 months

SECONDARY OUTCOMES:
Find a correlation between recurrence of supraventricular tachycardia and plasmatic aldosterone level before cardioversion | 6 months
Find a correlation between recurrence of supraventricular tachycardia and plasmatic ngal level before cardioversion | 6 months
Find a correlation between recurrence of supraventricular tachycardia and plasmatic galectin-3 level before cardioversion | 6 months
Find a correlation between recurrence of supraventricular tachycardia and occurrence of cardiovascular events | 6 months
Find a correlation between recurrence of supraventricular tachycardia and occurrence of renal failure | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: Yes